CLINICAL TRIAL: NCT04015206
Title: Effectiveness of Interpersonal Psychotherapy Group (IPT-G) as an add-on Strategy in the Treatment of Major Depression
Brief Title: Effectiveness of IPT-G in Major Depression
Acronym: IPT-GinMD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We completed One group intervention but the COVID Pandemic forced us to pause the research. We have preliminary data from 18 participants.
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0547
Record Dates: First submitted 2019-04-13; First posted 2019-07-10 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; Group Interpersonal Psychotherapy (IPT-G)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Study Type: Interventional Enrollment: 104 participants Allocation: Randomized Intervention Model: Parallel
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will aply the scales being blind for the arm the participant was assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPT-G+UCT (Experimental): 10 sessions of Group Interpersonal therapy added to pharmacotherapy + clinical management plus one individual session pre-group and one session pos-group
  Interventions: Other: Group Interpersonal Psychotherapy
- Usual treatment (UCT) (Active Comparator): Pharmacotherapy + Clinical management once a month
  Interventions: Other: Group Interpersonal Psychotherapy

INTERVENTIONS:
Other: Group Interpersonal Psychotherapy — Group Interpersonal Psychotherapy added to usual treatment (Pharmacotherapy + clinical management)
  Other Names: IPT-G

SUMMARY:
Although antidepressants are the primary treatment for major depression, response and remission rates are unsatisfactory. The primary objective of this study is to identify if adding interpersonal group therapy (IPT-G) to the usual psychopharmacological and clinical management treatment will improve depressive symptoms in major depression outpatients.

DETAILED DESCRIPTION:
Patients presenting a current unipolar depression episode (BDI-II > 18) without response to 2 adequate antidepressants trials (optimized by dose and time) will be randomly allocated to two arms: a) Treatment-as-usual (TAU) arm: antidepressant + Clinical management; b) Add-on strategy arm: 14 sessions of IPT-Group added to TAU.

IPT-Group will be delivered following manualized guidelines (WHO, 2016 and Stuart et al. 2012). The choice of antidepressants for TAU will be based on the Canadian Network for Mood and Anxiety Treatments (CANMAT) recommendations. Clinical management will follow the National Institute for Mental Health (NIMH) recommendations for clinical management.

Depression episode will be diagnosed using the Mini International Neuropsychiatric Interview (MINI-PLUS).

The following variables will be evaluated at baseline and the end of the add-on intervention in both arms of the study:

a) depression symptoms- Beck Depression Inventory (BDI-II; b) anxiety symptoms - Beck Anxiety Inventory (BAI); c) quality of life- World Health Organization Quality of life Instrument short version (WHOQOL-bref); d) social support- Medical Outcomes Study Social. Support Survey (MOS-SSS); e) resilience- The Brief Resilience Scale (BRS); f) attachment- The Adult Attachment Scale (AAS-R) Depression symptoms are the primary outcome. Anxiety symptoms and quality of life the secondary outcomes. Social support, resilience, and attachment will be considered as both secondary outcome and mediator or moderators in a multivariate model.

The database will be built using REDCap (Research Electronic Data Capture). Sample size estimation to detect a 5-point difference between the groups with a standard deviation of 6, considering α = 0,05 and power of 90%, suggests a 64 subjects sample. With the estimation of a loss of 25% of the sample during the study, 80 patients will be included (40 in each arm). A trained psychotherapist will conduct five IPT-G groups with eight patients in each group.

Study design and analysis will use Intention-to-treat analysis. For quantitative variables testing, student-T test t (normal distribution) or Mann Whitney (absence of normal distribution) will be used with a 5% level of significance. Categorical variables will be tested using the Chi-square with exact Fischer test with a 5% level of significance. Hierarchical linear regression will be used to determine the variables that could predict a reduction in the depression scores of the BDI-II. All analysis will be performed using the Statistical Package for the Social Sciences (SPSS) version 20.0.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Major Depressive Episode evaluated by the MINI-plus instrument.
2. Patients attending the depression outpatient clinic (HCPorto Alegre) for 6 months or more
3. History of two previous appropriate antidepressant treatments (dose: equivalent of 75 mg / day of amitriptyline and time: the minimum of four weeks)
4. Beck Depression Inventory scores above 18.

Exclusion Criteria:

1. Patients with bipolar disorder
2. Patients with substance abuse disorder,
3. Patients with risk of suicide
4. Patients with antisocial personality disorder
5. Patients with psychotic syndrome,
6. Patients with intellectual disability
7. Patients receiving some kind of psychotherapy at the present time and in the last four weeks.
8. Patients who are unable to communicate.
9. Patients with Dismissive Attachment Style

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-08-25 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Rate of Depression symptoms | 14 weeks
  The Beck Depression Inventory (BDI- II) brazilian version is an self-evaluation instrument, that the scale total scores aims to identify and quantify mild, moderate and severe depression. The patient is invited to answer how he has felt in the last week.
  The scale consists in 21 items including symptoms and attitudes, whose intensity varies from 0 to 3. The items refer to sadness, pessimism, past failure, lack of satisfaction, loss of pleasure, feelings of guilt, sense of punishment, self-steam, self-criticism, thoughts or desires of suicide, crying, agitation, loss of interest, indecision, devaluation, lack of energy, change in sleep patterns, irritability, changes in appetite, concentration difficulty, fatigue, loss of interest in sex.
  For patients diagnosed with Major Depression, the cut points are: 0-13 minimum, 14-19 mild depression, 20-28 moderate depression, 29-63 severe depression.

SECONDARY OUTCOMES:
Rate of Anxiety symptoms | 14 weeks
  The Beck Anxiety Inventory (BAI) brazilian version is a self-evaluation scale, total scores consists in 21 questions about how the individual has felt in the last week, expressed in common anxiety symptoms, such as sweating and feelings of anguish. The possible answers are: no, slightly, moderately and severely. The scores are: 0-10 minimum degree of anxiety, 11-19 mild anxiety, 20-30 moderate anxiety, 31-63 severe anxiety.
Rate of Quality of life domains | 14 weeks
  Differences in the World Health Organization Quality of life abbreviated questionaire instrument (WHOQOL-Bref) brazilian version scale scores in four domains (Physical, Psychological, Social Relationships and Environmental).
  Consists in 26 questions (each with a scale of Likert type composed of five degrees of intensity), two of them related to overall quality of life and health status and 24 facets of quality of life in general. The results can be: needs to improve (1 to 2,9), regular (3 to 3,9), good (4 to 4,9) and very good (5).
Rate of Social support | 14 weeks
  Difference in the Social Support Scale (MOS) validated for Brazil scores. Composed of self-applied items, multiple choice with a score of 1 to 5 (Likert scale) evaluates the perception of individuals on social support in health contexts. It consists in 19 items distributed in 4 dimensions: positive social interaction, possible social support, affective social support, emotional social support and informational social support. The patient should answer to each option: never, rarely, sometimes, often or always. In the end, the results are transformed in a punctuation of 0 to 100.
Rate of Resilience | 14 weeks
  Difference in the Brief Resilience Scale (BRS) total scores. The self-evaluation scale is a short version validated for Portuguese in Brazil and it is composed of 14 items, in the Likert format, with the score 1 to 7 for each question. It evaluates the perception of individuals about psychological characteristics linked to resilience. Higher overall scores indicate greater resilience. It is organized in 6 factors: self perception, future planning, social competences, family cohesion, social resources and structured style.
Style of Attachment | 14 weeks
  Difference in the Adult Attachment Scale (AAS-R) scores. The Portuguese version will be used, which has previously been used in the Brazilian population. It is a self-evaluation scale that consists in 18 items, marked on a Likert scale of 5 points. It measures the attachment style of the adults defined according to 3 dimensions: anxiety, comfort with proximity and confidence in others.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Fleck, PhD, Md., Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No